CLINICAL TRIAL: NCT04869046
Title: Intraoperative Wound Instillation of Levobupivacaine is Effective in Postoperative Pain Management for Hernia Repair in Children: a Randomized Controlled Clinical Trial
Brief Title: Levobupivacaine and Postoperative Pain Relief
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mother and Child Health Institute of Serbia Dr Vukan Cupic (Other)
Responsible Party: Principal Investigator, Maja Sujica MD MS, Maja Sujica, Head of Department of Anesthesiology and Intensive Care, Mother and Child Health Institute of Serbia Dr Vukan Cupic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4042/2
Record Dates: First submitted 2020-02-03; First posted 2021-05-03 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain; Inguinal Hernia Unilateral
Keywords: postoperative pain; hernia; children; levobupivacaine; instillation
MeSH Terms: conditions — Pain, Postoperative; Hernia | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levobupivacaine group (Experimental): Instillation of 0,1 ml/kg (0,5 mg/kg) levobupivacaine 0,5% in surgical wound before fascia closure
  Interventions: Drug: Instillation of levobupivacaine in surgical wound
- Control Group (Placebo Comparator): Instillation of 0,1 ml/kg 0,9% Sodium Chloride in surgical wound before fascia closure
  Interventions: Drug: Instillation of levobupivacaine in surgical wound

INTERVENTIONS:
Drug: Instillation of levobupivacaine in surgical wound — Once the hernia tissue had been surgically managed, the wound was sutured in layers and a solution of 0.5% levobupivacaine, 0.5 mg/kg (0.1 ml/kg), was instilled into the wound of children in the experimental group before suturing of the abdominal fascia. That same amount of 0.9% saline was given to children in the control group. The absorption of the solution took approximately 3 minutes, after which the wound was sutured. After completion of wound suturing, all children received 20 mg/kg of paracetamol administered as a rectal suppository.
  Other Names: Enteral analgesic mixture acetaminophen 10 mg/kg and ibuprofen 5mg/kg if needed; Acetaminophen, Ibuprofen

SUMMARY:
The study analysed direct levobupivacaine instillation in surgical wound and its effectiveness in postoperative pain control. Half participants received 0,5 % levobupivacaine and the other half received 0,9% saline solution

DETAILED DESCRIPTION:
Inguinal hernia is one of the most common conditions that requires elective surgical repair in children. The issue of post-operative pain in children is important, particularly because the surgical intervention per se is a stressful experience, after which the level of stressors in the recovery period should be minimized. Stress, including the pain in the postoperative period, could contribute to a delayed postoperative wound healing and recovery. Also, untreated acute pain could interfere with cognitive function, immune response as well as lead to the development of chronic postsurgical pain. For this reason, it is vital to reduce the painful sensations over the postoperative period as much as possible.

Levobupivacaine is a long-acting local anesthetic. Evidence from animal models and human volunteer participants showed that levobupivacaine has favourable effects on cardiovascular and central nervous systems. Clinical studies have also showed that levobupivacaine has a very low risk of systemic toxicity. A combination of levobupivacaine with non-opioid analgesics could have a beneficial role in the postoperative recovery from inguinal hernia surgery in terms of pain relief. The purpose of this study was to examine the effectiveness of levobupivacaine instillation combined with the routine postoperative non-opioid analgesia in children who underwent inguinal hernia repair.

It is very important for children to leave the hospital without additional support. Instilled levobupivacaine applied directly to the wound, currently interrupting transmission of the painful stimuli from the site of major trauma. The dose of applied levobupivacaine in this study is 2 times lower than that administered for caudal block and 4 times lower than the maximum dose. Analgesic effectiveness of this procedure is measured by the frequency of administration of a mixture of ibuprofen and acetaminophen over 24 hours after surgery, and duration of time between the administration of two doses.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery
* not having incarcerated hernia
* not having previous surgeries requiring general anaesthesia American Society of Anesthesia scores I and II
* not having allergy to topical anesthetics, paracetamol, ibuprofen and/or general anesthetics, opioids or muscle relaxants

Exclusion Criteria:

* worsening of health status prior to surgery
* parental withdrawal to study

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain assessment | "Min 30" if no changes "Hour 6"
  Assessment of pain by Face, Legs, Activity, Cry Consolability scale (nurse is observer) regularly, around the clock, first time 30 minutes after surgery, than after every 6 hours, until 24 h after surgery. Each score higher than 3 is considered significant and and an analgesic was given
Analgesic efficacy of nonopioid analgesic mixture | as needed in 24 hours
  30 minutes after taking analgesic mixture, the Face, Legs, Activity, Cry Consolability pain scale assessment was performed. Each score higher than 3 is considered significant and planed nonopioid analgesic was given. Frequency of nonsteroidal anti-inflammatory drug administration needed in 24 hour timeframe and time interval between doses were used as a measure of the analgesic effectiveness

SECONDARY OUTCOMES:
Control of breakthrough pain | as needed in 24 hours
  Breakthrough pain was treated with the same analgesic, in the same dose. The total allowed daily dose is taken into account. If it is exceeded, a dose of planned opioid analgesic is administered

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Vuckovic, MD, PhD, Study Director — University of Belgrade Faculty of Medicine
Locations (2):
- Serbia (2):
  - Institut for Mother and Child HealthCare "Dr Vukan Cupic", Belgrade
  - Institute for Mother and Child Health Care Dr Vukan Cupic, Belgrade

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams G, Howard RF, Liossi C. Persistent postsurgical pain in children and young people: prediction, prevention, and management. Pain Rep. 2017 Aug 21;2(5):e616. doi: 10.1097/PR9.0000000000000616. eCollection 2017 Sep. PMID 29392231
- [Background] Matsota P, Papageorgiou-Brousta M, Kostopanagiotou G. Wound infiltration with levobupivacaine: an alternative method of postoperative pain relief after inguinal hernia repair in children. Eur J Pediatr Surg. 2007 Aug;17(4):270-4. doi: 10.1055/s-2007-965473. PMID 17806025
- [Background] Dogra N, Dadheech R, Dhaka M, Gupta A. A study to compare caudal levobupivacaine, tramadol and a combination of both in paediatric inguinal hernia surgeries. Indian J Anaesth. 2018 May;62(5):359-365. doi: 10.4103/ija.IJA_747_17. PMID 29910493